CLINICAL TRIAL: NCT01026220
Title: A Non-Randomized Phase III Study of Response Adapted Therapy for the Treatment of Children With Newly Diagnosed High Risk Hodgkin Lymphoma
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Young Patients With Newly Diagnosed Hodgkin Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHOD0831; NCI-2011-01994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000660550; AHOD0831 (Other: Children's Oncology Group); AHOD0831 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-12

CONDITIONS: Childhood Nodular Lymphocyte Predominant Hodgkin Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage IV Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Vincristine; Vinorelbine; Cyclophosphamide; etoposide phosphate; Prednisone; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; indolepropanol phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Regimen I (consolidation therapy) (Experimental): Patients receive 2 more courses of ABVE-PC comprising doxorubicin hydrochloride IV over 1-120 minutes and cyclophosphamide IV over 30-60 minutes on days 1 and 2; bleomycin sulfate IV over at least 10 minutes or subcutaneously (SC) and vincristine sulfate IV on days 1 and 8; etoposide IV over 1-2 hours on days 1-3; oral prednisone twice daily on days 1-7; and filgrastim SC or IV daily beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: bleomycin sulfate; Drug: doxorubicin hydrochloride; Drug: liposomal vincristine sulfate; Drug: cyclophosphamide; Drug: etoposide phosphate; Drug: prednisone; Biological: filgrastim
- Regimen II (consolidation therapy) (Experimental): Patients receive ifosfamide IV continuously on days 1-4, vinorelbine ditartrate IV over 6-10 minutes on days 1 and 5, and filgrastim SC or IV beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity or disease progression. Patients then receive 2 more courses of ABVE-PC in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: bleomycin sulfate; Drug: doxorubicin hydrochloride; Drug: liposomal vincristine sulfate; Drug: vinorelbine tartrate; Drug: cyclophosphamide; Drug: etoposide phosphate; Drug: prednisone; Biological: filgrastim; Drug: ifosfamide
- Induction: all patient (Experimental): All patients receive ABVE-PC induction therapy then they are assigned to Group 2 (RER), Group 3 (SER) or taken off study if they develop progressive disease.
  Interventions: Drug: doxorubicin hydrochloride; Drug: liposomal vincristine sulfate; Drug: cyclophosphamide; Drug: etoposide phosphate; Drug: prednisone; Biological: filgrastim

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV or SC
  Other Names: Blenoxane; BLEO; BLM
  Arms: Regimen I (consolidation therapy); Regimen II (consolidation therapy)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: liposomal vincristine sulfate — Given IV
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
  Arms: Regimen II (consolidation therapy)
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide phosphate — Given IV
  Other Names: ETOP; Etopophos
Drug: prednisone — Given IV
  Other Names: DeCortin; Deltra
Biological: filgrastim — Given IV or SC
  Other Names: G-CSF; Neupogen
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
  Arms: Regimen II (consolidation therapy)

SUMMARY:
This phase III trial is studying how well giving combination chemotherapy together with radiation therapy works in treating young patients with newly diagnosed Hodgkin lymphoma. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill cancer cells. Giving combination chemotherapy together with radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To maintain the overall survival (as defined by 4-year "second-event" free survival) for subjects with high risk Hodgkin lymphoma at or above 95%.

SECONDARY OBJECTIVES:

I. To maintain 3-year event-free survival for subjects with high risk Hodgkin lymphoma at or above 93%.

II. To maintain comparable overall survival (as defined by 4-year "second-event" free survival) between subjects with high risk Hodgkin lymphoma who have a rapid or slow response to the initial 2 cycles of ABVE-PC* by intensifying therapy through the addition of 2 cycles of ifosfamide/vinorelbine in those with a slow early response.

III. To investigate whether very early response assessment measured by FDG-PET after 1 cycle of chemotherapy identifies a subject cohort that can be studied in future trials and that is distinguishable from currently defined RER after 2 cycles.

IV. To describe the patterns of relapse after ABVE-PC* and risk-adapted radiotherapy.

OUTLINE: This is a multicenter study.

INDUCTION THERAPY (ABVE-PC): Patients receive doxorubicin hydrochloride IV over 1-120 minutes and cyclophosphamide IV over 30-60 minutes on days 1 and 2, bleomycin sulfate IV over at least 10 minutes or subcutaneously (SC) and vincristine sulfate IV on days 1 and 8, etoposide phosphate IV over 1-2 hours on days 1-3, oral prednisone twice daily on days 1-7, and filgrastim* SC or IV daily beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity or disease progression.

NOTE: *Patients do not receive filgrastim on day 8.

Patients undergo clinical restaging and response assessment after 2 courses of induction therapy. Patients with rapid early response (RER) or slow early response (SER) proceed to consolidation therapy. Patients with progressive disease go off study.

CONSOLIDATION THERAPY: Patients are assigned to 1 of 2 consolidation therapy regimens based on response to induction therapy. Patients who develop progressive disease after induction are taken off protocol therapy.

REGIMEN I (RER): Patients receive 2 more courses of ABVE-PC in the absence of unacceptable toxicity or disease progression.

REGIMEN II (SER): Patients receive ifosfamide IV continuously on days 1-4, vinorelbine ditartrate IV over 6-30 minutes on days 1 and 5, and filgrastim SC or IV daily beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity or disease progression. Patients then receive 2 more courses of ABVE-PC in the absence of unacceptable toxicity or disease progression.

Patients with a continued response after completion of consolidation therapy proceed to risk-adapted radiotherapy.

RISK-ADAPTED RADIOTHERAPY: Beginning at 3 weeks after completion of consolidation chemotherapy, patients undergo radiotherapy once daily, 5 days a week, for 3 weeks (14 fractions) in the absence of unacceptable toxicity or disease progression. Patients classified as RER receive radiation therapy only to sites of bulky disease. Patients classified as SER receive radiation therapy to sites of bulky disease and areas that remain FDG-PET avid after induction therapy.

After completion of study therapy, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed newly diagnosed Hodgkin lymphoma (HL) meeting one of the following criteria:

  * Classical disease
  * Nodular lymphocyte-predominant disease
* Stage III or IV disease with B symptoms, as defined by ≥ 1 of the following:

  * Unexplained weight loss > 10% within the past 6 months
  * Unexplained recurrent fever > 38°C within the past month
  * Recurrent drenching night sweats within the past month
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR maximum serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 to 5 months)
  * 0.5 mg/dL (6 to 11 months)
  * 0.6 mg/dL (12 to 23 months)
  * 0.8 mg/dL (2 to 5 years)
  * 1 mg/dL (6 to 9 years)
  * 1.2 mg/dL (10 to 12 years)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (13 to 15 years)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (≥ 16 years)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* Shortening fraction ≥ 27% by ECHO OR ejection fraction ≥ 50% by MUGA (unless due to large mediastinal mass from HL)
* FEV_1/FVC > 60% by pulmonary function tests (PFT) (unless due to large mediastinal mass fromHL)

  * For children who are unable to cooperate for PFTs, the criteria are:

    * No evidence of dyspnea at rest
    * No exercise intolerance
    * Pulse oximetry > 92% on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pathologic prolongation of QTc interval (> 450 milliseconds) on 12-lead ECG
* No prior chemotherapy, biological response modifiers (e.g., monoclonal antibody therapy), or radiotherapy
* At least 28 days since prior corticosteroids except for emergent treatment for respiratory distress or spinal cord compression, or for treatment of allergy to contrast agent required for CT scan
* No other concurrent cancer chemotherapy or immunomodulating agents (including steroids)

  * Concurrent corticosteroid therapy as treatment or prophylaxis for anaphylactic reactions allowed
* No concurrent pegfilgrastim

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Kelly, MD, Principal Investigator — Children's Oncology Group
Locations (177):
- United States (156):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Vermont, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Israel (2):
  - Schneider Children's Medical Center of Israel, Petah Tikua
  - Chaim Sheba Medical Center, Tel Litwinsky
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Tie X, Shin M, Lee C, Perlman SB, Huemann Z, Weisman AJ, Castellino SM, Kelly KM, McCarten KM, Alazraki AL, Hu J, Cho SY, Bradshaw TJ. Automatic Quantification of Serial PET/CT Images for Pediatric Hodgkin Lymphoma Using a Longitudinally Aware Segmentation Network. Radiol Artif Intell. 2025 May;7(3):e240229. doi: 10.1148/ryai.240229. PMID 39969278
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- INDUCTION THERAPY (ABVE-PC): All Patients
- REGIMEN I (RER): Patients receive 2 more courses of ABVE-PC in the absence of unacceptable toxicity or disease progression.
- REGIMEN II (SER): Patients receive ifosfamide IV continuously on days 1-4, vinorelbine ditartrate IV over 6-30 minutes on days 1 and 5, and filgrastim SC or IV daily beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity or disease progression. Patients then receive 2 more courses of ABVE-PC in the absence of unacceptable toxicity or disease progression.
Period: Induction
Arm/Group | INDUCTION THERAPY (ABVE-PC) | REGIMEN I (RER) | REGIMEN II (SER)
Started | 166 | 0 | 0
Completed | 141 | 0 | 0
Not Completed | 25 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Physician Decision | 12 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0
Period: Consolidation Maintenance
Arm/Group | INDUCTION THERAPY (ABVE-PC) | REGIMEN I (RER) | REGIMEN II (SER)
Started | 0 | 81 | 80
Completed | 0 | 75 | 66
Not Completed | 0 | 6 | 14
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Arm/Group | INDUCTION THERAPY (ABVE-PC)
Number analyzed (Participants) | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 156
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 15 [5 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 112
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  Canada | 19
  United States | 143
  Australia | 3
  Puerto Rico | 1

OUTCOME MEASURES:

1. Primary Outcome: Second-event-free Survival
Description: Second event here is defined as any relapse/progression of Hodgkin Lymphoma (HL) or a previously reported second malignant neoplasm (SMN), a new SMN, or death after a first event which can be relapse/progression of HL, SMN, biopsy-proven HL following completion of Consolidation for Slow Early Response (SER) patient, positive bilateral bone marrow biopsy following completion of Consolidation for Stage IV patient, or death. If death occurs as the 1st event, it also counts as the 2nd event.
Time Frame: At 4 years from enrollment
Population: This analysis excludes n=20 patients who had protocol early terminations or deviations (n=4 Regimen I, n=12 Regimen II, and n=4 Induction only).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 1: All Patients
Arm/Group | Group 1
Number analyzed (Participants) | 145
Probability of survival | 0.91 [0.85 to 0.95]

2. Primary Outcome: Safety Analysis and Monitoring of Toxic Death
Description: The primary endpoint for safety analysis and monitoring is toxic death, which is death primarily attributable to treatment.
Time Frame: Within 30 days of protocol treatment at median follow-up of 48 months (range: 1 to 70 months).
Population: The six patients who received induction and reported death. The analysis here examines whether their death is primarily attributable to treatment or not.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: Event Free Survival
Description: Survival from enrollment to first event: relapse/progression, second malignancy, or death.
Time Frame: At 3 years from enrollment
Population: 164 Group 1 All Patients received induction therapy.
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Group 1
Number analyzed (Participants) | 164
Probability of survival | 0.81 [0.74 to 0.86]

4. Secondary Outcome: Second-event-free Survival
Description: as for outcome 1
Time Frame: At 4 years from enrollment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 2: Regimen 1
- Group 3: Regimen II
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 77 | 68
Probability of survival | 0.94 [0.84 to 0.98] | 0.88 [0.77 to 0.94]

5. Secondary Outcome: Event-free Survival for Rapid Early Response (RER) Positron Emission Tomography(PET)-1 Positive, RER PET-1 Negative
Description: To investigate whether very early response assessment measured by Fluorodeoxyglucose-PET after 1 cycle of chemotherapy identifies a subject cohort that can be studied in future trials and that is distinguishable from currently defined RER after 2 cycles.
Time Frame: 3 years from enrollment
Population: RER with positive PET-1, Event-Free Survival for RER PET-1 positive patients is compared to that of RER with negative PET-1: n=57 PET-1 positive RER patients, compared to 2 events among n=20 PET-1 negative RER patients. Two PET-1 equivocal RER patients (1 with relapse and 1 censored) are not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 4: RER PET-1 positive
- Group 5: RER PET-1 negative
Arm/Group | Group 1 | Group 4 | Group 5
Number analyzed (Participants) | 77 | 57 | 20
Probability of survival | 0.84 [0.73 to 0.91] | 0.82 [0.69 to 0.90] | 0.90 [0.65 to 0.97]

6. Secondary Outcome: Relapse-free Survival
Description: A description, survival to relapse, of patterns of relapse after Doxorubicin, Bleomycin, Vincristine, Etoposide - Prednisone, Cyclophosphamide (ABVE-PC) and risk-adapted radiotherapy.
Time Frame: 3 years from enrollment
Population: 161 patients began consolidation therapy: 126 patients received risk-adapted radiotherapy after consolidation therapy ABVE-PC and 35 did not.
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 6: risk-adapted radiation therapy
- Group 7: no risk-adapted radiation therapy
Arm/Group | Group 1 | Group 6 | Group 7
Number analyzed (Participants) | 161 | 126 | 35
Probability of survival | 0.82 [0.75 to 0.87] | 0.83 [0.75 to 0.88] | 0.79 [0.60 to 0.89]

7. Secondary Outcome: Event Free Survival
Description: Survival from enrollment to first event: relapse/progression, second malignancy, or death.
Time Frame: At 3 years from enrollment
Population: 161 patients began consolidation therapy: 81 Group 2 Regimen I and 80 Group 3 Regimen II.
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 2: Regimen I
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 81 | 80
Probability of survival | 0.83 [0.73 to 0.90] | 0.78 [0.67 to 0.86]

8. Secondary Outcome: Grade 3 and 4 Non-hematologic Toxicities During Protocol Therapy
Description: The number of patients that experience Common Terminology Criteria (CTC) Version 4 grade 3 or higher non-hematologic toxicity at any time during protocol therapy.
Time Frame: During and after completion of study treatment.
Population: 165 eligible patients.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 165
participants | 72

9. Secondary Outcome: Overall Survival
Description: Survival from enrollment to death.
Time Frame: At 3 years from enrollment
Population: 164 Group 1 All Patients received induction therapy. 161 patients began consolidation therapy: 81 Group 2 Regimen I and 80 Group 3 Regimen II.
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 164 | 81 | 80
Probability of survival | 0.97 [0.93 to 0.99] | 0.97 [0.90 to 0.99] | 0.97 [0.89 to 0.99]

ADVERSE EVENTS:
Description: Group 1 includes all patients and the Adverse Event reports of all events across the treatment procedure. Patients who experienced induction only are also included in Group 1. After induction patients were assigned to Group 2 (RER) and Group 3 (SER). While Group 2 and Group 3 are mutually exclusive, they are subsets of Group 1. Hence the Adverse Events in Group 1 will have overlaps with Adverse Events in Group 2 and Group 3.
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 89/165 | 43/81 | 46/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=165) | Group 2 (N=81) | Group 3 (N=80)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 39 (39) | 17 (17) | 22 (22)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 21 (21) | 12 (12) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 3 (3)
Oral pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 6 (6) | 3 (3) | 3 (3)
Flu like symptoms (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (5) | 5 (5) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 8 (8) | 2 (2) | 6 (6)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Upper respiratory infection (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 2 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 2 (2) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.